CLINICAL TRIAL: NCT04163042
Title: Physical Activity Counselling for Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Jennifer Brunet, Associate professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190643-01H
Record Dates: First submitted 2019-11-05; First posted 2019-11-14 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Survivorship; Cancer
Keywords: Physical activity; Behavioural support; Oncology; Telehealth; Self-determination theory; Behaviour change techniques; Young adult cancer survivors
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Videoconferencing intervention (Experimental): Participants allocated to group A will receive a behavioural support intervention via real-time videoconferencing.
  Interventions: Behavioral: 12-week videoconferencing behavioural support intervention to promote physical activity behaviour
- Group B: Usual care (No Intervention): Participants allocated to group B will receive usual care and will be advised to continue with their regular activities of daily living.

INTERVENTIONS:
Behavioral: 12-week videoconferencing behavioural support intervention to promote physical activity behaviour — Participants in Group A will receive six real-time, 1-on-1 60-minute sessions led by a physical activity counsellor over a 12-week period. Sessions will be delivered via videoconferencing and will aim to provide young adult cancer survivors with support as well as the knowledge, skills, and confidence to identify and overcome challenges to engaging in physical activity in order to increase physical activity behaviour and enhance patient-reported outcomes.
  Arms: Group A: Videoconferencing intervention

SUMMARY:
Survival rates for cancer are increasing, resulting in more young adult cancer survivors living with lingering side effects. Physical activity has been shown to improve the quality and length of life in young adult cancer survivors; yet, few are active enough, and little is currently being done to promote physical activity in this population. The investigators developed a novel behaviour support intervention to promote physical activity in young adult cancer survivors. In this two-arm pilot randomized controlled trial, the investigators aim to: (1) assess trial and intervention feasibility, (2) assess trial and intervention acceptability, and (3) generate data on physical activity behaviour. Young adult cancer survivors will be randomized to receive either a 12-week behaviour support intervention delivered via videoconferencing or will be allocated to usual care.

DETAILED DESCRIPTION:
Background: Young adults commonly experience persistent side effects following cancer treatment that impair quality of life. Physical activity (PA) holds promise as an intervention to mitigate persistent side effects and improve quality of life. Yet, few young adults are active enough to incur these benefits and efforts to promote PA following cancer treatment are lacking. Therefore, the investigators developed a novel behaviour support intervention to promote PA in young adults following cancer treatment, and have undertaken a pilot randomized controlled trial (RCT) to determine whether the intervention delivered via videoconferencing is both feasible and acceptable. Specifically, the aims of this ongoing parallel group two-arm pilot RCT are to: (1) assess trial and intervention feasibility and acceptability, and (2) generate data on PA behaviour.

Methods: Young adults who have completed cancer treatment are recruited from across Canada. Recruits are randomized to the intervention group (IG; i.e., a 12-week behaviour support intervention delivered via videoconferencing) or usual care (UC; no intervention). Drawing on the CONSORT 2010 statement and flow diagram, several feasibility outcomes pertaining to enrolment, allocation, follow-up, and analysis are tracked by study staff. Acceptability is assessed through interviews exploring IG and UC participants' experiences, thoughts, and perspectives of the trial, IG participants' views of the intervention and its mode of delivery, and PA counsellors' experiences delivering the intervention. PA is measured using accelerometers. Assessments take place at baseline (pre-randomization), post-intervention period, and at follow-up (24 weeks post-baseline).

Discussion: Feasibility and acceptability data will help determine if/what changes/modifications are needed to improve the trial protocol and/or intervention, and will inform the timeline for a definitive RCT. The PA behaviour data collected will inform sample size calculation for a future RCT that aims to test the effects of this intervention in young adults following cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Currently between the ages of 18-39 years;
* Received a first diagnosis of invasive cancer between the ages of 18-39 years;
* Completed primary treatment for cancer <5 years;
* Able to provide informed consent in English or French;
* Have approval of a healthcare provider to participate in the trial;
* Have access to videoconferencing technology (e.g., Skype, Google Hangouts, FaceTime).

Exclusion Criteria:

* Have evidence of current cancer (recurrent or secondary cancer or relapse);
* Currently meeting the Canadian Society for Exercise Physiology aerobic physical activity guidelines for cancer survivors in the month prior to enrolment (i.e., 150 minutes/week of moderate-to-vigorous intensity aerobic physical activity);
* Are non-ambulatory.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Duration of study (24 months)
  The number of eligible participants who enrol in the trial out of the number who are referred
Adherence rates | Duration of study (24 months)
  The number of intervention sessions attended out of the total recommended as part of the intervention
Acceptability of the trial and intervention | At week 12
  Participants will be asked to share their experiences, thoughts, and perspectives of the trial, the physical activity counsellor and the intervention by responding to open and close-ended questions during a semi-structured interview. Responses to close-ended questions will range from 1 ('poor' or 'not satisfied at all') to 10 ('excellent' or 'extremely satisfied').
Retention rates | Duration of study (24 months)
  The number of participants completing all three scheduled assessments.
Data completeness: Quantitative measures | Duration of study (24 months)
  The percentage of missing data on quantitative measures.
Data completeness: Qualitative interviews | Duration of study (24 months)
  The number of participants completing the acceptability interview following the intervention.

SECONDARY OUTCOMES:
Physical activity behaviour: 7-day accelerometer wear (objective physical activity behaviour) | Baseline (week 0), post-intervention (week 12), post-intervention follow-up (week 24)
  Change in participants' objective levels of physical activity as measured by accelerometers (ActiGraph GT3X+), which will be worn for a 7-day period across baseline (week 0), post-intervention (week 12), and follow-up (week 24).
Health-related quality of life: RAND 36-Item Short Form Health Survey (SF-36; Ware & Sherbourne, 1992) | Baseline (week 0), post-intervention (week 12), post-intervention follow-up (week 24)
  Change in participants' self-reported health-related quality of life across baseline (week 0), post-intervention (week 12) and post-intervention follow-up (week 24). The SF-36 measures eight dimensions: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Each item is scored on a 0 to 100 scale, with higher scores representing a more favourable health state.
Positive and negative affect: Positive and Negative Affect Schedule (PANAS-SF; Watson, Clark & Tellegen, 1998) | Baseline (week 0), post-intervention (week 12), post-intervention follow-up (week 24)
  Change in participants' self-reported positive and negative affect across baseline (week 0), post-intervention (week 12) and post-intervention follow-up (week 24). Each item is scored on a scale from 1 ('Very slightly or not at all') to 5 ('Extremely'). Items in the positive scale are averaged together to create a Positive Affect Score, and items in the negative scale are averaged together to create a Negative Affect Score. Higher positive and negative scores represent higher positive and negative affect, respectively.
Depressive symptoms: Patient Health Questionnaire Depression Scale (PHQ-9; Kroenke, Spitzer & Williams, 2001) | Baseline (week 0), post-intervention (week 12), post-intervention follow-up (week 24)
  Change in participants self-reported depressive symptoms across baseline (week 0), post-intervention (week 12) and post-intervention follow-up (week 24). Each item is scored on a 0 ('Not at all') to 3 ('Nearly every day') scale with higher scores representing greater severity of depressive symptoms.
Anxiety symptoms: 7-item Patient Health Questionnaire Generalized Anxiety Disorder Scale (GAD-7; Kroenke, Spitzer & Williams, 2006) | Baseline (week 0), post-intervention (week 12), post-intervention follow-up (week 24)
  Change in participants self-reported anxiety symptoms across baseline (week 0), post-intervention (week 12) and post-intervention follow-up (week 24). Each item is scored on a 0 ('Not at all') to 3 ('Nearly every day') scale, with higher scores representing greater severity of anxiety symptoms.
Impact of cancer: Impact of Cancer Instrument - Adolescent and Young Adult Module (Husson & Zebrack, 2017) | Baseline (week 0), post-intervention (week 12), post-intervention follow-up (week 24)
  Change in participants' self-reported perceptions of cancer impact from baseline (week 0), post-intervention (week 12) and post-intervention follow-up (week 24). Each item is scored on a scale from 0 ('Strongly disagree') to 4 ('Strongly agree'), with higher scores representing greater impact of cancer.
Motivation for physical activity: Behavioural Regulation in Exercise Questionnaire-3 (BREQ-3; Markland & Tobin, 2004) | Baseline (week 0), post-intervention (week 12), post-intervention follow-up (week 24)
  Change in participants' self-reported motivation for physical activity across baseline (week 0), post-intervention (week 12) and post-intervention follow-up (week 24). This measure taps six behavioural regulations in the physical activity context: amotivation, external, introjected, identified, integrated, and intrinsic motivation. Each item is scored on a scale from 0 ('Not true for me') to 4 ('Very true for me'), with higher scores reflecting greater amotivation, external, introjected, identified, integrated, and intrinsic motivation for physical activity.
Basic psychological need satisfaction in relation to physical activity: Psychological Need Satisfaction in Exercise Scale (PNSE; Wilson, Rogers & Rodgers, 2006) | Baseline (week 0), post-intervention (week 12), post-intervention follow-up (week 24)
  Change in participants self-reported psychological need satisfaction in relation to physical activity across baseline (week 0), post-intervention (week 12) and post-intervention follow-up (week 24). The PNSE measures perceptions of competence, autonomy and relatedness in relation to physical activity. Each item is scored on a scale from 1 ('False') to 6 ('True'), with higher scores representing greater perceived competence, autonomy and relatedness.
Autonomy support, structure and interpersonal involvement: Health Care Climate Questionnaire (Marcus et al., 1992) | Post-intervention (week 12)
  Participants perceived sense of autonomy support, structure and interpersonal involvement for physical activity post-intervention (week 12). Each item is scored on a scale from 1 ('Strongly disagree') to 7 ('Strongly agree'), with higher scores representing greater perceived autonomy support, structure and interpersonal involvement for physical activity.

OTHER OUTCOMES:
Socio-Demographic and Medical Information Questionnaire | Baseline (week 0)
  Self-reported socio-demographic and medical information (e.g., age, gender, civil and educational status, ethnicity) will be collected and used to describe the sample. Participants will be provided with a range of response options for each item.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Husson O, Zebrack BJ. Psychometric Evaluation of an Adolescent and Young Adult Module of the Impact of Cancer Instrument. J Adolesc Young Adult Oncol. 2017 Mar;6(1):159-170. doi: 10.1089/jayao.2016.0038. Epub 2016 Sep 21. PMID 27654343
- [Background] Marcus BH, Rakowski W, Rossi JS. Assessing motivational readiness and decision making for exercise. Health Psychol. 1992;11(4):257-61. doi: 10.1037//0278-6133.11.4.257. PMID 1396494
- [Derived] Brunet J, Price J, Gillison F, Standage M, Taljaard M, Beauchamp MR, Reed J, Srikanthan A. Feasibility and acceptability of a parallel, two-arm randomized controlled trial to evaluate an online physical activity behavior counseling intervention for young adults diagnosed with cancer: a mixed-methods pilot study. Pilot Feasibility Stud. 2025 Nov 4;11(1):131. doi: 10.1186/s40814-025-01701-w. PMID 41189005
- [Derived] Brunet J, Price J, Srikanthan A, Gillison F, Standage M, Taljaard M, Beauchamp MR, Reed J, Wurz A. The physicAl aCtivity Counselling for young adult cancEr SurvivorS (ACCESS) trial: A protocol for a parallel, two-arm pilot randomized controlled trial. PLoS One. 2022 Dec 30;17(12):e0273045. doi: 10.1371/journal.pone.0273045. eCollection 2022. PMID 36584027
- See also: Psychological Need Satisfaction in Exercise Scale — https://doi.org/10.1123/jsep.28.3.231
- See also: Behavioural Regulation in Exercise Questionnaire-3 — https://doi.org/10.3389/fpsyg.2018.01940